CLINICAL TRIAL: NCT04497285
Title: HOPE: Real World Clinical Practice Study to Assess the Impact of Using Comprehensive Genomic Data on the Next Treatment Decision Making Choice in Patients With Locally Advanced or Metastatic Breast Cancer in Spain
Brief Title: Real World Study Using Comprehensive Genomic Data on the Next Treatment Decision Making in Metastatic Breast Cancer
Acronym: HOPE
Status: Active, not recruiting | Type: Observational
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry); Roche Pharma AG (Industry); Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SOLTI-1903
Record Dates: First submitted 2020-07-03; First posted 2020-08-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample collection and collection of tumor tissue block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: blood sample collection and collection of tumor tissue block — blood sample collection and collection of tumor tissue block

SUMMARY:
SOLTI 1903 HOPE is a national, real world clinical practice study conducted in patients diagnosed with metastatic breast cancer who are receiving, have just received or will receive treatment for its advanced disease. Patients will lead their inclusion, participation and follow-up in the study through a digital tool, but they are encouraged to include their physician's in this study. Tissue samples from metastatic (preferred) or primary tumor will be collected for analyses, together with blood samples. A Molecular Advisory Board (MAB) will assess and give recommendations according patient's molecular profile.

The primary objective is to assess the real-world clinical practice of integration of molecular profiling in the Standard of Care (SoC) management of mBC patients connected through a digital tool.

DETAILED DESCRIPTION:
Eligible patients are those who are 18 or older, either female or male, confirmed locally advanced or metastatic breast cancer of any subtype and who have received, are receiving, or will receive any line of treatment from metastatic disease.

Demographic data, disease characteristics, treatment history, and quality of life data will be collected through a digital tool by the patient. The data are de-identified and will be used to advance multiple areas of research into mBC. The study will be complemented by a patient empowerment program that will include informative workshops and video-tutorials about precision medicine and the HOPE study itself. Tumor tissue samples must be submitted for genomic profiling using FoundationOne CDx. Blood samples for circulating tumor DNA (ctDNA) profiling using Guardant360 also will be collected.

Molecular reports will be reviewed by the Molecular Advisory Board (MAB) and recommendations according to the molecular profile will be sent to the patients and physicians through the digital tool to let them know these treatment options and also notified about clinical trials for which they may be eligible.

The primary objective is to assess the real-world clinical practice of integration of molecular profiling in the Standard of Care (SoC) management of mBC patients connected through a digital tool. Secondary objectives include: to describe genetic mutational profile from both tests, to evaluate if a patient-centric strategy could achieve better enrollment than the classical approach site-physician-patient, and to assess the efficacy of the program to allocate patients in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients.
2. Age ≥18 years.
3. Signed informed consent prior to any screening procedure.
4. Locally advanced or metastatic breast cancer of any subtype confirmed both pathologically and radiologically (stage IIIb- IV disease).
5. The subjects must be about to receive, or receiving, or will have completed treatment for their metastatic disease with any line of treatment in either a clinical trial or the healthcare setting.
6. Availability of one metastatic (preferably), primary tumor sample or blood sample.
7. Measurable or non-measurable disease.
8. Quality of life score according to ECOG scale ≤ 3.
9. Minimal life expectancy of 6 months.

Exclusion Criteria:

1. Inability to consent or conform to the processes involved in a clinical study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic breas cancer
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Metastatic breast cancer management based on tumor molecular profile | 1 year after end of accrual
  The number of patients assigned to different treatments based on the genomic profile.

SECONDARY OUTCOMES:
Description of the genetic mutational profile in tumor tissue. | Ongoing basis during 3 years' patient recruitment
  To describe the genetic mutational profile of the patients using Foundation One CDx.
Description of the genetic mutational profile in blood samples | Ongoing basis during 3 years' patient recruitment
  To describe the genetic mutational profile of the patients using liquid biopsy (Guardant360 test).
Description of the enrollment rate of the study | Ongoing basis during 3 years' patient recruitment
  To describe the enrollment rate using the HOPE patient centric strategy (videotutorials and user experience of different technologies as the digital tool).
Feasibility of implementing the program for metastatic breast cancer | 1 year after end of accrual and subsequently during follow up period of 5 years
  To describe number of patients who are allocated to clinical trials and number of patients allocated on on-label therapies considering tumor genomic profile.
Correlation between efficacy endpoints among patients enrolled in clinical trials according to the tumor's genomic profile and among patients receiving SoC. | 1 year after end of accrual and subsequently during follow up period of 5 years
  To describe of PFS and OS among the patients enrolled in clinical trials according to the tumor's genomic profile, and among the patients receiving SoC.
Quality of life assessment using EuroQol-5D (EQ-5D) in patients with metastatic breast cancer | Ongoing basis during 3 years' patient recruitment
  The EuroQol EQ-5D is designed to assess health status in terms of a single index value or utility score. It contains 5 descriptors of current health state (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having 5 levels of function (1=no problem, 2=slight problem, 3=moderate problem, 4=severe problem, and 5=unable/extreme). The scores on the 5 descriptors are summarized to create a single summary score. The EQ-5D also includes a visual analog scale (VAS), in which the patients self-rate their overall health status on a scale from 0 (worst imaginable) to 100 (best imaginable).
Quality of life assessment using Functional Assessment of Cancer Therapy FACT-B in patients with metastatic breast cancer | Ongoing basis during 3 years' patient recruitment
  The FACT-B consists of the Functional Assessment of Cancer Therapy-General (FACT-G) (27-items) and a breast-specific module: a 10-item instrument designed to assess patient concernsrelating to BC. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Patients are asked to respond to a Likert scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.

CONTACTS AND LOCATIONS:
Locations (1):
- Translational Genomics and Targeted Therapeutics in Solid Tumours Lab in August Pi i Sunyer Biomedical Research Institute (IDIBAPS), Barcelona, Please Select, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olivera-Salguero R, Segui E, Cejalvo JM, Oliveira M, Tolosa P, Vidal M, Malumbres M, Gavila J, Saura C, Pernas S, Lopez R, Margeli M, Balmana J, Munoz M, Blancas I, Boni V, Ciruelos E, Galve E, Perello A, Sanchez-Bayona R, de la Cruz S, de la Hoya M, Galvan P, Sanfeliu E, Gonzalez-Farre B, Sirenko V, Blanch-Torras A, Canes J, Masanas H, Olmos R, Forns M, Prat A, Casas A, Pascual T. HOPE (SOLTI-1903) breast cancer study: real-world, patient-centric, clinical practice study to assess the impact of genomic data on next treatment decision-choice in patients with locally advanced or metastatic breast cancer. Front Oncol. 2023 Apr 28;13:1151496. doi: 10.3389/fonc.2023.1151496. eCollection 2023. PMID 37188177